CLINICAL TRIAL: NCT06453876
Title: Percutaneous Embolectomy, Ultrasund Assisted Low Dose Thrombolysis or Heparin for Intermediate High Risk Pulmonary Embolism
Brief Title: Percutaneous Embolectomy, Ultrasound Assisted Thrombolysis or Heparin for Intermediate High Risk Pulmonary Embolism
Acronym: STRATIFY-II
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jesper Kjaergaard (Other)
Collaborators: Zealand University Hospital (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor-Investigator, Jesper Kjaergaard, Consultant MD PhD DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRATIFY-II 1.0 (04OCT2023)
Record Dates: First submitted 2023-12-04; First posted 2024-06-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Heparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomized allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Unfractionated Heparin / Low molecular heparin and thrombolysis if needed (Active Comparator): Standard medical Therapy for intermediate-high risk pulmonary embolism
  Interventions: Drug: Heparin
- Ultrasound assisted Thrombolysis (Active Comparator): Ultrasound assisted Thrombolysis using teh EKOS system. 10 mg af alteplase over 6 hours total and heparin
  Interventions: Device: Ultrasound assisted Thrombolysis
- Percutaneous Thrombectomy (Active Comparator): Percutaneous Embolectomy using the Inari (R) Flowtriever thrombectomy system (R) and heparin
  Interventions: Device: Percutaneous Embolectomy

INTERVENTIONS:
Device: Ultrasound assisted Thrombolysis — Please see Arms
  Other Names: EKOS system
  Arms: Ultrasound assisted Thrombolysis
Device: Percutaneous Embolectomy — Please see arms
  Other Names: Inari FlowTriever
  Arms: Percutaneous Thrombectomy
Drug: Heparin — Active comparator
  Other Names: Unfractionated or low molecular weight heparin
  Arms: Unfractionated Heparin / Low molecular heparin and thrombolysis if needed

SUMMARY:
The STRATIFY II trial investigates the efficacy of three different approaches to reducing thrombus burdon in patients with acute intermediate high-risk pulmonary embolism: percutaneous embolectomy (the Flow Triever® system, INARI medical), USAT (EKOS® system, Boston Scientific with low dose alteplase) and heparin with the option to perform full-dose thrombolysis. As a co-primary secondary end point the trial assess the incremental efficacy of the embolectomy vs the catheter based low dose thrombolysis approach.

Thus the two main hypothesis being tested are:

1. Thrombus burden reduction after 48-96 h is increased with a catheter based (embolectomy or USAT) compared to the a heparin with optional high dose thrombolysis approach (1st co-primary outcome)
2. Thrombus burden reduction after 48-96 h is increased with percutaneous embolectomy compared to USAT with low-dose alteplase (2nd co-primary outcome)

DETAILED DESCRIPTION:
BACKGROUND Intermediate high-risk PE is associated with an up to 10% risk of death even if the circulations of the patient is only marginally impacted (1). Full dose thrombolysis has been investigated is two randomized trials but finding the intervention to be efficacious in preventing hemodynamic deterioration, but at the cost of an increased risk og bleeding with cancels the benefit of thrombolysis with regards to risk of death (2, 3). Therefore recent guidelines suggest that patients are managed by heparins with thrombolysis available as a rescue therapy if the patient deteriorates hemodynamically (1). Further two small clinical have trials have investigated the role of low dose thrombolysis finding a substantial reduction in late incidence of pulmonary hypertension (4) and similar efficacy of half dose thrombolysis and lower occurrence of bleeding compared to full doses thrombolysis (5).

Since then catheter based interventions for administering low Thrombolysis for acute PE has been introduced. Some interventionalists use simple catheters while the EKOS® system of USAT claims to increase the efficacy of thrombolytics by applying a mechanical force from ultrasound emitting crystals nead the emboli while slowly administering the thrombolytics near the thrombus in the pulmonary arteries. The USAT techniques has been tested in a small randomized trial, finding the treatment to efficacious in terms of reducing right heart dilatation (6). Later a dose finding RCT should similar efficacy of dosages of alteplase in USAT ranging from 4 mg to 24 mg per catheter (7). The HI-PEITHO trial (NCT04790370) is a 406 patient trial current enrolling patients, and the STRATIFY trial from our group (NCT04088292) is a 210 patient trial also currently including patients, and thus more knowledge of the efficacy of this approach will be available in 1-2 years.

Recently catheter-based embolectomy has been introduced. While no randomized trials have compared this technique to the guidelines supported strategy of UFH or LMWH, several registries and sace series have been put forward, suggesting a significant efficacy and a acceptable risk of bleeding. The INARI FlowTriever system ® has been use in a substantial number of patients, but have only been reported in none peer-reviewed presentation as results of two registries comparing patients treated with percutaneous embolectomy and a registry describing 'real world data' has been presented online (8) and in comment section in medical journals (9). An ongoing randomized trial comparing percutaneous embolectomy and catheter directed thrombolysis, is currently recruiting patients (NCT05111613)(10) and another comparing embolectomy and heparins is planned (NCT06055920).

Balancing the risk and efficacy of the treatment strategy remains important and since a lack of data both proving the efficacy of the novel treatment alternatives and limited data comparing efficacy in trial with a suitable design, a clinical equipoise remains.

TRIAL OBJECTIVES AND HYPOTHESIS The STRATIFY II trial investigates the efficacy of three different approaches to reducing thrombus burdon in patients with acute intermediate high-risk pulmonary embolism: percutaneous embolectomy (the Flow Triever® system, INARI medical), USAT (EKOS® system, Boston Scientific with low dose alteplase) and heparin with the option to perform full-dose thrombolysis. As a co-primary secondary end point the trial assess the incremental efficacy of the embolectomy vs the catheter based low dose thrombolysis approach.

Thus the two main hypothesis being tested are:

1. Thrombus burden reduction after 48-96 h is increased with a catheter based (embolectomy or USAT) compared to the a heparin with optional high dose thrombolysis approach (1st co-primary outcome)
2. Thrombus burden reduction after 48-96 h is increased with percutaneous embolectomy compared to USAT with low-dose alteplase (2nd co-primary outcome) SETTING AND PATIENT POPULATION SETTING The trial is including patients diagnosed with an acute PE (defined as symptom duration of less than 14 days) with intermediate- high risk , please see section of definition below. Patients are recruited from participating centers by the attending cardiologist, either in the emergency room or at the ward. Since risk stratification most often involves a cardiologist the investigators expect the majority of patients to be included in the trial immediately after risk stratification.

The participants will be informed on the possible inclusion in the trial in the ward, and every measure possible will be taken to ensure a quit environment for the information. The patient will be informed about their right to have an assessor present during the information session, and that they may take the time needed to consider their participation in the trial and giving their informed consent. The informed consent will be obtained soon after the patient have been informed on their diagnosis of intermediate-high risk PE.

DEFINITIONS Definition of Intermedidate- high risk PE is based on ESC guideline classification from 2019 (1) as identification of PE in the pulmonary main trunk, main and segmental pulmonary arteries on CT angiography performed as part of the diagnostic work-up of patients with clinical suspicion of acute PE RV dysfunction is defined as

* RV/LV ratio of > 1 on CT angiography or echocardiography (apical 4 chamber view in-diastole) OR
* RV systolic function by visual assessment or TAPSE < 18 mm OR
* TR gradient > 40 mmHg Elevated Cardiac Biomarker
* Increase in cardiac Troponins (I or T) above normal OR
* Increase Creatine Kinase MB (CKMB) above normal OR
* Increase in NT-pro-BNP above normal In the absence of shock at time of screening defined as
* Systolic blood pressure > 100 mmHg INCLUSION CRITERIA

  1. Age ≥ 18 years
  2. Informed consent for trial participation
  3. Intermediate high-risk PE according to ESC criteria
  4. Thrombus visible in main, lobar or segmental pulmonary arteries on CT angiography
  5. 14 days of symptoms or less EXCLUSION CRITERIA

  <!-- -->

  1. Altered mental state (GCS < 14)
  2. No qualifying CT angiography performed (> 24 hour since CT angiography)
  3. Females of child bearing potential, unless negative HCG test is present
  4. Thrombolysis for PE within 14 days of randomization
  5. Thrombus passing through patent Foramen Ovale (risk of paradoxical embolism)
  6. Ongoing oral anticoagulation therapy (heparins, aspirin, antiplatelet therapy and NOAC allowed)
  7. Comorbidity making 6 months survival unlikely
  8. Absolute contraindications for thrombolysis

     1. Hemorrhagic stroke or stroke of unknown origin at any time
     2. Ischemic stroke in the preceding 6 months
     3. Central nervous system damage or neoplasms
     4. Recent major trauma/surgery/head injury in the preceding 3 weeks
     5. Gastrointestinal bleeding within the last month
     6. Known bleeding risk Relative contraindications do not preclude randomization. Relative contraindications include: Transient ischemic attack in the preceding 6 months, Oral anticoagulant therapy, Pregnancy, or within one week post partum, Non-compressible puncture site, Traumatic resuscitation, Refractory hypertension (systolic blood pressure >180 mm Hg), Advanced liver disease, Infective endocarditis, Active peptic ulcer OUTCOMES CO-PRIMARY ENDPOINT
* Reduction in modified Miller score (score of thrombus involvement and segmental flow)(11, 12) comparing percutaneous treated groups (embolectomy and USAT combined) to heparin/LMWH group, p<0.01 (n=140 vs. n=70).
* Reduction in modified Miller score (score of thrombus involvement and segmental flow)(11, 12) comparing percutaneous embolectomy and USAT, p<0.04 (n=70 vs n=70) SECONDARY ENDPOINTS
* • Bleeding complications (major and minor bleeding complication according to the Thrombolysis in Myocardial Infarction classification)
* Duration of index admission, including hospital-based rehabilitation
* Dyspnoea index (Visual analogue scale) after 48-96 h and after 3 months
* FiO2, blood pressure, and respiratory rate, heart rate at time of follow-up CTPA
* Mortality in the three groups (log-rank), and hazard ratio in multivariable analysis using the UFH/LMWH as a reference
* Incidence of TR gradient > 40 mmHg at 3 months follow-up echocardiography
* 6MWT at 3 months follow up comparing the three groups
* Quality of life at 3 months follow-up comparing the three groups (PEmb-Qol and 5Q-5D-5L)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Informed consent for trial participation
3. Intermediate high-risk PE according to ESC criteria
4. Thrombus visible in main, lobar or segmental pulmonary arteries on CT angiography
5. 14 days of symptoms or less

Exclusion Criteria:

1. Altered mental state (GCS < 14)
2. No qualifying CT angiography performed (> 24 hour since CT angiography)
3. Females of child bearing potential, unless negative HCG test is present
4. Thrombolysis for PE within 14 days of randomization
5. Thrombus passing through patent Foramen Ovale (risk of paradoxical embolism)
6. Ongoing oral anticoagulation therapy (heparins, aspirin, antiplatelet therapy and NOAC allowed)
7. Comorbidity making 6 months survival unlikely
8. Absolute contraindications for thrombolysis

   1. Hemorrhagic stroke or stroke of unknown origin at any time
   2. Ischemic stroke in the preceding 6 months
   3. Central nervous system damage or neoplasms
   4. Recent major trauma/surgery/head injury in the preceding 3 weeks
   5. Gastrointestinal bleeding within the last month
   6. Known bleeding risk Relative contraindications do not preclude randomization. Relative contraindications include: Transient ischemic attack in the preceding 6 months, Oral anticoagulant therapy, Pregnancy, or within one week post partum, Non-compressible puncture site, Traumatic resuscitation, Refractory hypertension (systolic blood pressure >180 mm Hg), Advanced liver disease, Infective endocarditis, Active peptic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-05 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Thrombus burdon reduction (intervention vs. heparin) | To end of inclusion + 96 hours
  Reduction in modified Miller score (score of thrombus involvement and segmental flow) comparing percutaneous treated groups (embolectomy and USAT combined) to heparin/LMWH group, p<0.01 (n=140 vs. n=70)
Thrombus burdon reduction (USAT vs. embolektomy) | To end of inclusion + 96 hours
  Reduction in modified Miller score (score of thrombus involvement and segmental flow) comparing percutaneous embolectomy and USAT, p<0.04 (n=70 vs n=70)

SECONDARY OUTCOMES:
Bleeding complications (major and minor bleeding complication according the TIMI classification) | 3 months
  TIMI classification
Duration of index admission, including hospital based rehabilitation | 3 months
  Duration of index admission
Dyspnea index (Visual analog scale) after 48-96 hours and after 3 months | 96 hours and 3 months
  Duration of index admission
Rate of further interventions for pulmonary embolism during index admission | 3 months
  (embolectomy, full dose thrombolysis, mechanical ventilation, need for vasopressors, cardio pulmonary resusuctation, VA-ECMO etc)
Mortality in the three groups (log-rank), and hazard ratio in multivariable analysis using the UFH/LMWH as reference. Inclusion date of last patient's 3 month follow-up defines last day of follow-up | 1 year on avarage, at least 3 months
  Clinical outcome
Incidence of TR gradient > 40 mmHg at 3 months follow-up echocardiography | through study completion, an average of 1 year
  Incidence of TR suggestive of pulmonary hypertension
6MWD at 3 months comparing the three groups | 3 months
  Functional test
Quality of life at 3 months follow-up comparing the three groups (PEmbQoL) | 3 months
  QoL

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital Gentofte, Gentofte Municipality, Capital Region
  - Copenhagen University Hospital Bispebjerg Hospital, Bispebjerg
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Copenhagen University Hospital, Herlev Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No